CLINICAL TRIAL: NCT01849354
Title: Operative Treatment of Endometriosis Patients in Turku University Hospital
Acronym: ProEndo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Carita Edgren, MD, Turku University Hospital
Other Study IDs: T17/2013
Record Dates: First submitted 2013-02-19; First posted 2013-05-08 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood and urine samples. Peritoneal fluid, helthy peritoneum, endometriosis tissue and endometrium samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Endometriosis patients: Endometriosis patients to be operated in Turku university hospital 2013-2015
- Control patients: Patients who will be operated because of an adnexal finding other than endometriosis, for example ovarian cyst. Also patients with laparoscopic sterilization will be recruited to the control group.

SUMMARY:
The women's clinic at Turku University Hospital has also since year 2000 accomplished and systematically increased advanced surgical treatment for the endometriosis patients with difficult disease. The aim is to centralize endometriosis treatment in the hospital district and by doing that be able to offer exact diagnosis, advanced surgical treatment and infertility treatment for every patient in the hospital area. The main purpose of this study is to find out how the operative treatment of endometriosis patients in Turku University Hospital is functioning and to see how the quality of life of these patients is before and after the surgery. Furthermore, the structure of the endometriosis patients' endometrium and the different markers of blood and urine are studied.

DETAILED DESCRIPTION:
This prospective study is performed with the women's clinic in Turku University Hospital.

The aim is to get every patient, who is operated because of endometriosis in Turku University Hospital, to participate on the study. The patients are recruited on the basis of the referral letters, which have been sent to the endometriosis outpatient clinic. Before the visit to the outpatient clinic they are sent an electric form in which it is told about the study and the samples to be collected and from the voluntariness of the participation and privacy protection. The patients fill in the electric anamnesis form, which is gone through with the outpatient clinic visit. With the outpatient clinic visit the patients sign a consent form together with the doctor. After having agreed to the study the patients will fill an electric questionnaire about quality of life of endometriosis patient (EHP-30) and a questionnaire about their sexual satisfaction (FSFI) before the operation. The electric forms are made on the Webropol-program. In the electric forms the patient information is encoded so that an individual patient cannot be identified.

The control group consists of patients who will be operated because of an adnexal finding other than endometriosis, for example ovarian cyst. Also patients with laparoscopic sterilization will be recruited to the control group. The patients who might be suitable, are contacted by telephone call. The main points of the study are explained to them and they are asked to participate in the study. The control patients fill in the same electric forms before the operation as the endometriosis patients do and doctor discusses with them before they agree to the study. The exclusion criterions are acute infection, pregnancy, hemoperitoneum, suspicion of a malignancy or incidentally found endometriosis.

The findings during the operation of endometriosis patients and the procedures that have been done are documented on the specific forms made for this purpose (Oper1, -2 ja -3-forms) and the prognostic form for future fertility (Endometriosis Fertility Index) is filled. On the morning of the operation day the urine and blood samples are taken and the samples from endometrium, peritoneum and peritoneal fluid as well as the endometriotic tissue are collected during the operation.

Blood and urine samples are taken also from the control patients on the morning of the operation day. During the operation the samples from peritoneum, peritoneal fluid and endometriotic tissue are collected.

After 4-6 months of the operation all the patients come to outpatient clinic visit to Turku University Hospital's women's clinic. Before this visit they fill in the specific electric questionnaire for the control visit. In this form they are asked for example how well they have recovered from the operation and how their symptoms have developed. They also fill in the EHP-30- and FSFI-forms. The endometrial and blood and urine samples are collected during this visit. After this all patients will receive an annual follow up form electrically 1, 2 and 3 years after the operation in which they are asked about later recovery, symptoms and possible pregnancies and the patients will also fill in the EHP-30- and FSFI-forms.

The information from the questionnaires is encoded so that an individual patient cannot be identified. The questionnaires and the register collected from them will be stored in Turku University Hospital at least until the study has ended.

ELIGIBILITY:
Inclusion Criteria:

* Endometriosis
* Adnexal finding
* Laparoscopic sterilization

Exclusion Criteria:

* Pregnancy
* Acute infection
* Hemoperitoneum
* Suspicion of a malignancy

Max Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Endometriosis patients to be operated in Turku university hospital 2013-2015. The control group consists of patients who will be operated because of an adnexal finding other than endometriosis, for example ovarian cyst. Also patients with laparoscopic sterilization will be recruited to the control group.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Endometriosis related pain symptoms before and after the endometriosis surgery | 3 years
  Endometriosis related pain symptoms are collected from the operativelly treated endometriosis patients by a questionnaire 6 months, 1, 2 and 3 years after the surgery by using NRS-scale.
The quality of life before and after the endometriosis surgery | 3 years
  Quality of life is assessed with EHP-30 questionnaire before and 6 months, 1, 2 and 3 years after the endometriosis surgery
Sexual functioning before and after endometriosis surgery | 3 years
  Sexual functioning is measured by using FSFI (Female Sexual Function Index)-form before, 6 months, 1, 2 and 3 years after endometriosis surgery.

SECONDARY OUTCOMES:
Novel diagnostic markers for endometriosis | 3 years
  Samples of blood, urine, endometrium and endometriosis tissue are collected during the operation and analyzed to find novel diagnostic markers for endometriosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland